CLINICAL TRIAL: NCT05889377
Title: Socket Preservation Technique Using Bovine Bone, Platelet Rich Fibrin Or A Combination Of Both: A Clinical, Radiographic And Histological Assesment At 4 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Christian Makary, Professor, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XFMD218
Record Dates: First submitted 2023-05-11; First posted 2023-06-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-05

CONDITIONS: Ridge Preservation; Post Extraction Alveolar Bone Resorption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bovine Bone (Experimental)
  Interventions: Procedure: Socket preservation
- Platelet Rich Fibrin (Experimental)
  Interventions: Procedure: Socket preservation
- Bovine Bone + PRF (Experimental)
  Interventions: Procedure: Socket preservation
- Control (No Intervention)

INTERVENTIONS:
Procedure: Socket preservation — Socket preservation will be done after tooth extraction. For each group we will use a bone substitute.
  Arms: Bovine Bone; Bovine Bone + PRF; Platelet Rich Fibrin

SUMMARY:
Post extraction alveolar bone resorption is one of the main challenges that face oral implantologists in their daily surgical practice (1). To palliate to post-extraction resorption, advanced bone grafting and regeneration techniques have been described (2). However, these procedures, although well documented and validated, still have relatively high complication rates and patient morbidity, in addition to the elevated cost and duration of treatment (3). Socket preservation is a very useful technique in order to counter post extraction resorption issues, therefore eliminating the need for future complicated and delicate regeneration procedures (4). Many biomaterials were proposed for socket preservation such as allografts and bovine hydroxyapatite (5). Recently autologous platelet concentrates such as Platelet Rich Fibrin PRF were described as a potential socket filler material (6).

In the proposed protocol, fresh extraction sockets will be either grafted by a bovine bone substitute, a PRF plug or a mixture of both. Sockets will then be clinically and radiographically monitored over time to assess three-dimensional soft and hard tissue stability. Bone quality will be histologically examined at 6 months implant placement. A no graft group will serve as control.

The results of this study may be of major importance since they could give an objective idea of the most efficient socket preservation technique, thus offering simple and secure oral rehabilitation solutions for both patient and practitioner.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will require single tooth extraction and subsequent implant rehabilitation.
2. Patients over 18 years of age.
3. Patients willing to comply with the study requirements (signed consent form)
4. Good oral hygiene and no signs of active periodontal infection
5. No compromising medical status
6. < 10 cigarettes smoking per day

Exclusion Criteria:

1. acute myocardial infarction within the last two months;
2. Uncontrolled coagulation disorders;
3. uncontrolled diabetes (HBA1c> 7.5);
4. radiation therapy to the head \ neck region in the last 24 months;
5. immunocompromised patients, HIV positive or receiving chemotherapy in the last five years;
6. past or present treatment with intravenous bisphosphonates;
7. psychological or psychiatric problems;
8. abuse of alcohol or drugs;

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Hard tissue change by measuring bone profil retraction between 0,4 and 12 months using 3D slicer software | 4 and 12 months
  Comparison of the bone profile change by CBCT dicom files superimposition at different time frame
Soft tissue change by measuring gingival retraction between 0,4 and 12 months using 3D slicer sftware | 4 and 12 months
  Comparison of the soft tissue profile change by STL files superimposition at different time frame

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided